CLINICAL TRIAL: NCT07056530
Title: Effectiveness of Telenursing in Improving Self-Care and Blood Pressure Control Among Adults With Chronic Hypertension: A Quasi-Experimental Study in Türkiye
Brief Title: Effectiveness of Telenursing on Self-Care and Blood Pressure Control in Adults With Hypertension
Acronym: TELENURSING-HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dursun Alper YILMAZ (Other)
Responsible Party: Sponsor-Investigator, Dursun Alper YILMAZ, Research Assistant, Agri Ibrahim Cecen University
Organization: Agri Ibrahim Cecen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TELENURSING-HTN-2025-AICU; 919B012319310 (Other: The Scientific and Technological Research Council of Turkey (TÜBİTAK))
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Nursing; Telenursing
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, non-randomized, parallel design comparing an 8-week telenursing intervention group to a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group received a structured telenursing program consisting of weekly phone-based counseling sessions for 8 weeks, focusing on medication adherence, healthy nutrition, physical activity, stress management, and blood pressure self-monitoring.
  Interventions: Behavioral: Telenursing Counseling
- Control Group (No Intervention): Participants in this group received usual care provided by the hospital without any additional telenursing counseling.

INTERVENTIONS:
Behavioral: Telenursing Counseling — Structured weekly phone-based counseling sessions delivered by a trained nurse for 8 weeks, focusing on medication adherence, healthy lifestyle behaviors, stress management, and self-monitoring of blood pressure.
  Other Names: Weekly Remote Nursing Counseling
  Arms: Intervention Group

SUMMARY:
This quasi-experimental study aims to evaluate the effectiveness of a structured telenursing program in improving self-care practices and blood pressure control among adults with chronic hypertension in Türkiye. Participants received weekly telephone-based nursing counseling for eight weeks, focusing on medication adherence, healthy nutrition, physical activity, stress management, and regular self-monitoring. The study compares changes in blood pressure and self-care scores between the intervention and control groups.

DETAILED DESCRIPTION:
Hypertension remains one of the most prevalent chronic diseases worldwide, significantly contributing to cardiovascular morbidity and mortality. Despite advances in pharmacological treatment, non-pharmacological support and patient self-care play a crucial role in achieving optimal blood pressure control. This study was designed as a quasi-experimental pretest-posttest controlled trial to test whether a structured telenursing intervention improves self-care behaviors and blood pressure outcomes in adults with chronic hypertension.

The study was conducted at Ağrı Training and Research Hospital in Türkiye between March 2024 and March 2025. A total of 151 participants aged 30-75 years were recruited and assigned to an intervention group or a control group. The intervention group received weekly telephone-based nursing counseling sessions delivered by trained nurses for eight consecutive weeks. Counseling covered key self-care topics including medication adherence, dietary modifications, physical activity, stress reduction, and blood pressure self-monitoring. The control group received usual care.

Primary outcomes included changes in systolic blood pressure and mean arterial pressure. Secondary outcomes included changes in self-efficacy and self-care practices measured by the Hypertension Self-Care Profile (HTN-SCP). Ethical approval was obtained from Ağrı İbrahim Çeçen University Scientific Research Ethics Committee (Approval No: E102912). Official permission for implementation was provided by the Ağrı Provincial Directorate of Health (Approval No: E24156). The study was supported by TÜBİTAK (Project No: 919B012319310). Findings from this study aim to support the use of telenursing as a cost-effective digital health strategy for chronic disease management in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic hypertension for at least 1 year.
* Aged between 30 and 75 years.
* Able to communicate via telephone.
* Provided informed consent to participate.

Exclusion Criteria:

* Diagnosed with severe comorbid conditions (e.g., advanced heart failure, cancer).
* Cognitive impairment that prevents communication.
* Hearing impairment that prevents phone counseling.
* Participation in another hypertension intervention program within the last 6 months.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) | Baseline and 8 weeks post-intervention
  Difference in mean systolic blood pressure from baseline to 8 weeks after the intervention.

SECONDARY OUTCOMES:
Change in Hypertension Self-Care Profile (HTN-SCP) Score | Baseline and 8 weeks post-intervention
  Difference in mean HTN-SCP score from baseline to 8 weeks post-intervention to assess improvement in self-care behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Dursun Alper Yılmaz, PhD, Study Chair — Ağrı İbrahim Çeçen Üniversitesi
Locations (1):
- Ağrı İbrahim Çeçen University, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset includes personal health information and no additional consent for public sharing was obtained. Only summary results will be published in scientific journals.